CLINICAL TRIAL: NCT02875587
Title: Cabergoline Versus Calcium Gluconate Infusion in the Prevention of Ovarian Hyperstimulation Syndrome. A Randomized Controlled Trial
Brief Title: Cabergoline Versus Calcium Gluconate Infusion in the Prevention of Ovarian Hyperstimulation Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Principal Investigator, Prof .Usama M.Fouda, M.D, PhD, Aljazeera Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Cabergoline/calcium gluconate
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: OHSS
Keywords: OHSS; Infertility; Cabergoline; Calcium gluconate; IVF-ET
MeSH Terms: conditions — Infertility | interventions — Cabergoline; Calcium Gluconate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cabergoline group (Active Comparator): Cabergoline is administered starting on the day of HCG administration.
  Interventions: Drug: Cabergoline
- Calcium gluconate infusion group (Experimental): Calcium gluconate is administered starting on the day of HCG administration.
  Interventions: Drug: Calcium gluconate

INTERVENTIONS:
Drug: Cabergoline — Cabergoline (Dostinex; Pfizer, Italy) at a daily dose of 0.5 mg is administered orally at bed time for 8 days starting on the day of HCG administration
  Arms: Cabergoline group
Drug: Calcium gluconate — Intravenous 10% calcium gluconate, 10 mL in 200 mL of physiologic saline on the day of ovum pickup, day 1, day 2, and day 3 after ovum pickup. Intravenous infusion will be performed within 30 minutes.
  Arms: Calcium gluconate infusion group

SUMMARY:
The aim of this study is to compare the efficacy of calcium gluconate infusion versus cabergoline in the prevention of ovarian hyperstimulation syndrome (OHSS) in patients pretreated with GnRH agonist long protocol who are at high risk for OHSS.

DETAILED DESCRIPTION:
Ovarian hyperstimulation syndrome (OHSS) is a serious complication of assisted reproduction.

Previous studies revealed that calcium gluconate infusion reduced the risk of OHSS. Other studies revealed that cabergoline (potent dopamine receptor agonist on D2 receptors)was effective in preventing OHSS.

The aim of this study is to compare the efficacy of calcium gluconate infusion versus cabergoline in the prevention of ovarian hyperstimulation syndrome (OHSS) in patients pretreated with GnRH agonist long protocol who are at high risk for OHSS.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are stimulated using the long luteal GnRH agonist protocol and at high risk for developing OHSS [have more than 18 follicles (> 11mm) and serum estradiol ≥ 3000 pg/ml on the day of HCG administration].

Exclusion Criteria:

* Fibrosis of lung
* Swelling or inflammation around the heart or lung
* Hypertension
* Liver disease
* Heart valve disease and allergy to cabergoline or ergot derivatives.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2016-10; Primary Completion 2018-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Moderate or severe ovarian hyperstimulation syndrome | Within 4 weeks of HCG adminstration

SECONDARY OUTCOMES:
The Number of Participants Who Achieved Ongoing Pregnancy | 18 weeks after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Usama M Fouda, M.D,PhD, Study Chair — Aljazeera( Al Gazeera) hospital
Locations (2):
- Egypt (2):
  - Aljazeera hospital, Giza
  - Riyadh Fertility and Reproductive Health center, Giza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gurgan T, Demirol A, Guven S, Benkhalifa M, Girgin B, Li TC. Intravenous calcium infusion as a novel preventive therapy of ovarian hyperstimulation syndrome for patients with polycystic ovarian syndrome. Fertil Steril. 2011 Jul;96(1):53-7. doi: 10.1016/j.fertnstert.2011.04.094. Epub 2011 May 31. PMID 21621772